CLINICAL TRIAL: NCT00172965
Title: Diagnosis of Oral Precancers and Cancers Using Optic Coherence Tomography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700341
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2004-08

CONDITIONS: Oral Cancers
Keywords: Optic coherence tomography; oral cancer; oral precancers
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Diagnosis of oral precancers and cancers using optic coherence tomography

DETAILED DESCRIPTION:
Diagnosis of oral precancers and cancers using optic coherence tomography

ELIGIBILITY:
Inclusion Criteria:

* oral cancer, oral precancers

Exclusion Criteria:

* other diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-08; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Pin Chiang, DMSc, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan